COSMOS: NCT NCT03035201 COSMOS-Mind: NCT102422745

# LA-Aging Summary Measures from Cognitive Assessment Battery April 11, 2023

#### **Global Cognitive Function Domain**

# GC1. General Cognitive Function

- Test: TICSm
- Variable: totalscore from TICS
- Approach
  - Create z-score by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation
  - Ignore any missing data

# **Memory Domain**

# MEM1. Word List Delayed Memory

- Test: TICSmApproach
  - Create z-score by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation
  - o Ignore any missing data

# MEM2. Story Memory Immediate

- Test: Story Recall
- Variable: totscore from storyrecall1; story packet
- Approach
  - Separately, for scores from each packet, create z-scores by dividing the difference between individual scores and the raw cohort-wide baseline mean by the raw cohortwide standard deviation
  - o Take mean of immediate recall scores for each participant
  - o Renormalize mean to have standard deviation 1
  - Ignore any missing data

# MEM3. Story Memory Delayed

- Test: Story Recall
- Variables: totscore from storyrecall2; story packet
- Approach
  - Separately, for scores from each packet, create z-scores by dividing the difference between individual scores and the raw cohort-wide baseline mean by the raw cohortwide standard deviation
  - Take mean of delayed recall scores for each participant
  - Renormalize mean to have standard deviation 1
  - o Ignore any missing data

## **Executive Function Domain**

#### EF1. Set shifting

- Test: OTMT-B
- Variables: time\_comp\_b
- Approach

COSMOS: NCT NCT03035201 COSMOS-Mind: NCT102422745

- Transform score by using a log transformation
- Create z-score by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation
- Re-order z-scores so that positive scores reflect better performance by subtracting each from 0
- Ignore any missing data

## EF2. Category Verbal Fluency

- Tests: Category and Letter Fluency
- Variables: animalcorrect; vegecorrect
- Approach for Category Verbal Fluency
  - Sum animal and verbal fluency scores (requires both to be non-missing)
  - Create z-score by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation

# **EF3.** Letter Verbal Fluency

- Variables: lcorrect; fcorrect
- Approach for Letter Fluency
  - Sum "I" and "f" scores (requires both to be non-missing)
  - Create z-score by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation

#### EF4. Attention/Working Memory 1

- Test: Number Span Forward and Backward
- Variables: dst\_forwardtot; dst\_backwardTot
- Approach
  - Sum digit forward and backwards scores (requires both to be non-missing)
  - Create z-scores by dividing the difference between individual scores and the raw cohortwide baseline mean by the raw cohort-wide standard deviation

#### **Composite Scores**

## **General Cognitive Function**

Equal to GC1

## Global Episodic Memory

- Average MEM1-MEM3, ignoring any missing data
- Create z-score by dividing the difference between individual scores and the raw cohort-wide baseline mean by the raw cohort-wide baseline standard deviation

#### **Global Executive Function**

- Average EF1-EF4, ignoring any missing data
- Create z-score by dividing the difference between individual scores and the raw cohort-wide baseline mean by the raw cohort-wide baseline standard deviation

#### **Global Cognitive Composite**

- Average z-scores from the following individual tests (note that this differs from averaging the three domain-specific z-scores and includes TICSm (Long) and Oral Trails A, which don't contribute to any of these):
  - TICSm total score
  - o TICSm-Long to assess delayed memory
  - Story recall (immediate)
  - Story recall (delayed)

COSMOS: NCT NCT03035201 COSMOS-Mind: NCT102422745

- Oral trails A (based on log transformation
- Oral trails B (based on log transformation)
- Verbal fluency
- Category fluency
- Number span test (total of forward and backward)
- Create z-score by dividing the difference between individual scores and the raw cohort-wide baseline mean by the raw cohort-wide standard deviation

In the primary analyses, to follow intention-to-treat and use all available data to compare changes from baseline, we will include all cognitive assessments (baseline through Year 3) as dependent variables in general linear models (including data from participants with incomplete follow-up) and use linear contrasts to compare the average changes from baseline across follow-up between intervention groups: the difference between the average means at years 1, 2, and 3 and the baseline mean.